CLINICAL TRIAL: NCT07101926
Title: Monitoring of Anti-TFPI in Hemophilia EUREKA
Brief Title: Monitoring of Anti-TFPI in Hemophilia
Acronym: EUREKA
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0342
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia; Rebalancing Agents; Prophylaxis
MeSH Terms: conditions — Hemophilia A | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The specific types of samples that will be retained include platelet-rich plasma (PRP) and platelet-poor plasma (PPP) derived from citrated whole blood.
  During a routine visit, four citrate tubes of 2.7 mL each (totaling 10.8 mL) will be collected per patient. PRP is prepared by centrifugation at 150 × g for 10 minutes at 18°C within 30 minutes of collection. The plasma is carefully transferred to avoid leukocyte contamination and adjusted to a standardized platelet count if necessary.
  These samples will be used for thrombin generation testing, specifically via the Calibrated Automated Thrombogram (CAT) method, and will not be stored for long-term use-no long-term storage is planned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe adult haemophilia A or B patient with factor levels ≤2%: * 6 on prophylaxis with FVIII or FIX concentrates after an adequate washout period of 48h for SHL FVIII molecules, at least 4 days for EHL-FVIII Fc and at least 10 days for EHL-FIX molecules
  * 5 receiving prophylaxis with marstacimab.
  Interventions: Biological: blood sampling

INTERVENTIONS:
Biological: blood sampling — One-time peripheral blood draw (10.8 mL total, 4 citrated tubes) collected during a routine clinical visit for thrombin generation testing on platelet-rich and platelet-poor plasma. No additional medical procedures or treatments are involved in the study.

SUMMARY:
During the development of anti-TFPI antibodies, thrombin generation assay (TGA) was employed using both in vitro measurements (antibodies added to blood samples) and ex vivo approaches (blood samples from patients in phase II and III trials). While a significant improvement in thrombin generation was observed in all samples from patients with severe hemophilia, no correlation with clinical outcomes could be established. Notably, thrombin peak levels were consistently improved even in patients who experienced bleeding episodes. These measurements were conducted in platelet-poor plasma (PPP) with standard reagents, which may not adequately reflect the hemostatic efficacy of anti-TFPI antibodies given their mechanism of action. It is hypothesized that optimizing reagents and utilizing more appropriate biological materials could enhance TGA sensitivity, as previously demonstrated for monitoring emicizumab.

The absence of a laboratory assay to monitor anti-TFPI (tissue factor pathway inhibitor) antibodies poses a significant challenge for managing patients in surgical settings and treating acute severe bleeding. This study aims to develop a reliable assay to evaluate the hemostatic efficacy of anti-TFPI antibodies and their combined procoagulant effect with factor concentrates (FVIII or FIX) or bypassing agents.

ELIGIBILITY:
* Inclusion Criteria :

  * - Male Patient
  * 18 years old
  * severe hemophilia patients A or B (FVIII < 1%,FIX<=2%)
  * on prophylaxis with FVIII or IX concentrates after an adequate washout period of 48h for SHL FVIII molecules, at least 4 days for EHL-FVIII Fc and at least 10 days for EHL-FIX molecules.
  * On prophylaxis with Marstacimab
  * Willing to participate
  * Capable of following protocol procedures under investigator appreciation
* Exclusion Criteria :

  * - patients refusing to provide 4 additional blood tubes for research
  * Patient with an other coagulation disorder
  * patients who received an injection of FVIII or FIX during the required washout period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentials patients for this study will be identified within the department of clinic hemostasis at Louis Pradel Hospital and Necker Hospital during their routine visit. Hemophila patients are coming regularly to the hospital for their consultaion and a blood drawn
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Development of a Laboratory Assay to Assess Hemostatic Efficacy of Anti-TFPI Antibodies | At time of sample analysis (single visit; Day 0)
  Assessment of the thrombin generation assay's ability to evaluate the procoagulant effect of anti-TFPI antibodies alone and in combination with factor concentrates (FVIII or FIX) or bypassing agents (rFVIIa, aPCC).

SECONDARY OUTCOMES:
Analytical Sensitivity of TGA to Anti-TFPI Antibodies | Day 0
  Evaluate the effect of different TGA conditions (e.g., low TF concentration, use of PRP, CTI) to enhance sensitivity to anti-TFPI antibodies.
Identification of Optimal TGA Parameters for Monitoring Anti-TFPI Effect | Day 0
  Determine which parameters (e.g., thrombin peak, ETP, lag time, velocity, time to peak) best reflect the action of anti-TFPI antibodies under optimized assay conditions.
Correlation Between TGA Parameters and Clinical Use of Anti-TFPI Therapies | Day 0
  Compare TGA results from 5 patients treated with marstacimab and 3 patients with concizumab to assess correlation with clinical treatment exposure.
Detection of Hypercoagulability from Combined Therapy in TGA | Day 0
  In vitro testing of anti-TFPI antibodies in combination with FVIII, FIX, rFVIIa, or aPCC to assess risk of excessive thrombin generation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupement hospitalier Est Hôpital Cardilogique Service d'hémostase clinique, Bron
  - Centre de Référence Hémophilie et autres déficits rares en protéine de la coagulationCentre de Traitemendes Hémophiles F. Josso, Paris

IPD SHARING:
Plan to Share IPD: Undecided